CLINICAL TRIAL: NCT02096393
Title: A Prospective, Randomised Control Trial Assessing Clinical and Radiological Outcomes of Patient Specific Instrumentation In Total Knee Arthroplasty
Brief Title: Patient Specific Instrumentation in TKR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STH16313
Record Dates: First submitted 2014-03-07; First posted 2014-03-26 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient specific instrumentation (Experimental): The patient will undergo using patient specific instrumentation
  Interventions: Device: Zimmer Patient specific instruments
- Standard instrumentation (Active Comparator): The patient will undergo surgery using standard instrumentation
  Interventions: Device: Standard instrumentation

INTERVENTIONS:
Device: Zimmer Patient specific instruments — A custom made cutting block will be used during total knee replacement surgery. The cutting block is made specific to patient's anatomy based on MRI scans taken 6 weeks prior to surgery.
  Arms: Patient specific instrumentation
Device: Standard instrumentation — Standard instrumentation will be used during total knee replacement surgery.
  Arms: Standard instrumentation

SUMMARY:
This is a randomised control trial to assess the benefits of using patient specific instrumentation in total knee replacement surgery. Patient specific instrumentation is an individualised system for total knee replacement surgery. The system has been marketed and is already in use in some centres. The type of implant used remains the same but the sizing of the components, and alignment of the implant is expected to improve. This study assesses any improvement in implant alignment in using the patient specific instrumentation, any improved intra-operative outcomes and any long term clinical outcome improvements for patients.

DETAILED DESCRIPTION:
This is a randomised control trial to assess the benefits of using patient specific instrumentation in total knee replacement surgery. Patient specific instrumentation is an individualised system for total knee replacement surgery. The system has been marketed and is already in use in some centres. The process is similar to traditional knee replacement surgery but approximately 6 weeks prior to the operation patients will undergo an MRI scan of their knee, hip and ankle. From this data the dimensions and rotation of the knee can be accurately measured, and a custom made jig can be made specific to that patients anatomy. The jig is used intra-operatively to make accurate bone cuts according to this pre-operative plan, the type of implant used remains the same but the sizing of the components, and alignment of the implant is expected to improve. This study assesses any improvement in implant alignment in using the patient specific instrumentation, any improved intra-operative outcomes and any long term clinical outcome improvements for patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-75 years at time of surgery.
* Those presenting with primary or secondary osteoarthritis and/or rheumatoid arthritis of the knee.
* Those deemed capable of giving informed consent, understanding the aims of the study and expressing willingness to comply with the post-operative review programme.
* Patients who signed the study consent form prior to surgery.

Exclusion Criteria:

* Pregnant women.
* Those whose prospects for a recovery to independent mobility would be compromised by known coexistent, medical problems.
* Those with a known co-existent medical condition where death is anticipated within five years due to the pre-existing medical condition.
* Previous knee surgery including those already treated by with a total knee replacement (i.e. requiring a revision knee replacement).
* Muscle contracture around the knee joint
* Individuals with active or suspected infection or sepsis.
* Patients with contraindication to MRI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Implant alignment | 6 weeks
  Sagittal and coronal alignment of the knee arthroplasty implant will be measured on full length radiographs

SECONDARY OUTCOMES:
Oxford Knee Score | 1yr, 5yr, 10yr
  Patient questionnaire

OTHER OUTCOMES:
EUROQOL-5D | 1 year, 5 years and 10 years
IKKS Score | 1yr, 5 yr, 10yr
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Blakey, MBChB, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Rotherham District General Hospitals NHS Trust, Rotherham, South Yorkshire
  - Sheffield Teaching Hospital NHS Trust, Sheffield, South Yorkshire